CLINICAL TRIAL: NCT02748148
Title: Implementing an Enhanced Standardized Medication Therapy Management Approach Within a Primary Care Setting
Brief Title: Implementation Study of Enhanced Medication Therapy Management in Primary Care Practice
Acronym: EMTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tabula Rasa HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MTM-309
Record Dates: First submitted 2016-04-01; First posted 2016-04-22 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Medication Therapy Management; Pharmacogenomics
Keywords: Medication Therapy Management; Pharmacogenomics
MeSH Terms: interventions — Medication Therapy Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medication therapy management (Experimental): Medication therapy management service that is enhanced by the incorporation of pharmacogenomics and medication risk mitigation factor technology
  Interventions: Other: Medication therapy management

INTERVENTIONS:
Other: Medication therapy management — Implementation of a systematic approach to evidence- and personalized-based medicine through a pharmacist-guided medication therapy management service
  Other Names: Enhanced medication therapy management

SUMMARY:
The purpose of this study is to identify challenges and successes associated with implementing an enhanced medication therapy management service in primary care practice.

DETAILED DESCRIPTION:
The specific aim of this study is to implement a Medication Therapy Management (MTM) service in primary care that is enhanced by the incorporation of pharmacogenomics (PGx) and medication risk mitigation (MRM) factor technology and is standardized by a systematic approach to evidence- and personalized-based medicine. The primary objective is to implement the systematic approach to delivering an enhanced MTM service in a primary care setting. Secondary objectives include: determine how successful the communication between prescriber and pharmacist is within implementing the service, determine how PGx testing can be incorporated into primary care prescribers' daily work flow, determine if patients are receptive to PGx testing, determine how satisfied prescribers are with an enhanced MTM clinical service and their confidence to conduct on their own, and determine if enhanced MTM optimizes or changes drug therapy for patients.

ELIGIBILITY:
Inclusion Criteria:

* Receiving primary health care from Elmwood Family Physicians; and
* Medicare beneficiary; and
* Currently prescribed at least 7 medications, or prescriber feels patient would benefit from enhanced medication therapy management, or actual or suspected medication-related problem

Exclusion Criteria:

* Not willing to participate in the study and sign informed consent; or
* Non-English speaking or designated surrogate as translator not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Qualitative description of process-related challenges and successes as assessed by observation and survey | 3 months
  Implementation

SECONDARY OUTCOMES:
Quantitative description of bidirectional communication as assessed by turn-around times from pharmacist's recommendations delivered to prescriber's responses received | 3 months
  Communication
Qualitative description of incorporation of pharmacogenomic testing into workflow and receptiveness as assessed by observation and survey | 3 months
  Pharmacogenomic testing
Qualitative description of prescriber satisfaction with enhanced medication therapy management services as assessed by survey | 3 months
  Prescriber survey
Qualitative and quantitative description of potential impact of enhanced medication therapy management services on drug regimens as assessed by before-and-after observations | 3 months
  Impact

CONTACTS AND LOCATIONS:
Overall Officials: Kevin T Bain, PharmD, MPH, Principal Investigator — Tabula Rasa HealthCare
Locations (1):
- Elmwood Family Physicians, Marlton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Budnitz DS, Shehab N, Kegler SR, Richards CL. Medication use leading to emergency department visits for adverse drug events in older adults. Ann Intern Med. 2007 Dec 4;147(11):755-65. doi: 10.7326/0003-4819-147-11-200712040-00006. PMID 18056659
- [Background] Kongkaew C, Noyce PR, Ashcroft DM. Hospital admissions associated with adverse drug reactions: a systematic review of prospective observational studies. Ann Pharmacother. 2008 Jul;42(7):1017-25. doi: 10.1345/aph.1L037. Epub 2008 Jul 1. PMID 18594048
- [Background] Classen DC, Pestotnik SL, Evans RS, Lloyd JF, Burke JP. Adverse drug events in hospitalized patients. Excess length of stay, extra costs, and attributable mortality. JAMA. 1997 Jan 22-29;277(4):301-6. PMID 9002492
- [Background] Ernst FR, Grizzle AJ. Drug-related morbidity and mortality: updating the cost-of-illness model. J Am Pharm Assoc (Wash). 2001 Mar-Apr;41(2):192-9. doi: 10.1016/s1086-5802(16)31229-3. PMID 11297331
- [Background] Evans WE, Relling MV. Pharmacogenomics: translating functional genomics into rational therapeutics. Science. 1999 Oct 15;286(5439):487-91. doi: 10.1126/science.286.5439.487. PMID 10521338
- [Background] Doan J, Zakrzewski-Jakubiak H, Roy J, Turgeon J, Tannenbaum C. Prevalence and risk of potential cytochrome P450-mediated drug-drug interactions in older hospitalized patients with polypharmacy. Ann Pharmacother. 2013 Mar;47(3):324-32. doi: 10.1345/aph.1R621. Epub 2013 Mar 12. PMID 23482734
- [Derived] Schwartz EJ, Turgeon J, Patel J, Patel P, Shah H, Issa AM, Knowlton OV, Knowlton CH, Bain KT. Implementation of a Standardized Medication Therapy Management Plus Approach within Primary Care. J Am Board Fam Med. 2017 Nov-Dec;30(6):701-714. doi: 10.3122/jabfm.2017.06.170145. PMID 29180545